CLINICAL TRIAL: NCT00847431
Title: Mapping Mood in the Subthalamic Nucleus in PD
Brief Title: Mapping Mood in the Subthalamic Nucleus in Parkinson's Disease (PD)
Acronym: MOOD-D
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08-0354; R01NS058797-05 (NIH)
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease; Depression; Anxiety
Keywords: Subthalamic Nucleus; Deep Brain Stimulation; Depression; Anxiety; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- STN DBS Group: PD patients with deep brain stimulators in the subthalamic nucleus. Subjects within this group will be placed into either a 1 contact group, or 2 contact group, depending on contact location requirements for this study.
- Control Group: PD patients without deep brain stimulator surgery, with similar symptoms to the study group.

SUMMARY:
The goal of this study is to determine the vulnerability of mood-related neurocircuitry in Parkinson Disease (PD) using deep brain stimulation of the subthalamic nucleus (STN DBS).

ELIGIBILITY:
Inclusion Criteria for STN-DBS subjects:

* Age 40 or older
* DBS STN Surgery in past 2 to 36 months
* Ability to tolerate turning off Stimulators
* Ability to read and comprehend questions
* English speaking

Exclusion Criteria for STN-DBS subjects:

* Other severe complications post surgery: stroke, seizure, major loss of consciousness, other brain trauma/surgery, or head injuries(i.e. near drowning), encephalitis, or hydrocephalus, blindness, deafness
* Clinically determined Dementia ( Most recent MMSE score of >24)

Inclusion Criteria for Control subject:

* Age 40 or older
* Ability to read and comprehend questions
* English speaking

Exclusion Criteria for Control subject:

* Other severe complications post surgery: stroke, seizure, major loss of consciousness, other brain trauma/surgery, or head injuries(i.e. near drowning), encephalitis, or hydrocephalus, blindness, deafness
* Clinically determined Dementia ( Most recent MMSE score of >24)
* Plans to have DBS STN surgery in the next 24 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients with and without STN DBS
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2008-12; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara G Hershey, PhD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - University of Cincinnati, Movement Disorder Center, Cincinnati, Ohio